CLINICAL TRIAL: NCT00510978
Title: One Year, Randomised, Double Blind, Placebo Controlled Trial of Probiotics, Bifidobacterium Infantis 35624 or Lactobacillus Salivarius UCC118, as Food Supplements for Maintenance of Remission in Crohn's Disease and Ulcerative Colitis
Brief Title: Probiotics in GastroIntestinal Disorders
Acronym: PROGID
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College Cork (Other)
Collaborators: European Commission (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CT900/301/1-2; QLK1-CT-2000-00563
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2007-08

CONDITIONS: Ulcerative Colitis; Crohn's Disease
Keywords: Inflammatory Bowel Disease IBD; Ulcerative Colitis; Crohn's disease; Probiotics; Gastrointestinal
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Bifidobacterium infantis 35624
  Interventions: Biological: Bifidobacterium infantis 35624
- 2 (Active Comparator): Lactobacillus salivarius UCC118
  Interventions: Biological: Lactobacillus salivarius UCC118
- 3 (Placebo Comparator): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Bifidobacterium infantis 35624 — 1 sachet/day for one year
  Arms: 1
Biological: Lactobacillus salivarius UCC118 — 1 sachet per day for 1 year
  Arms: 2
Biological: Placebo — 1 sachet per day for 1 year
  Arms: 3

SUMMARY:
All of us have millions of bacteria living in our gut. These bacteria are very important to our health providing us with protection against infections of the gut, allowing us to gain extra nutritional value from food we eat and helping our immune system. Changes in the balance of these many bacteria can make us vulnerable to infections both from within and from outside the gut. Certain bacteria may also be directly associated with some diseases of the gut. Research by doctors and scientists into relationships between the bacteria normally found in our gut and certain diseases of the gut is helping to develop food supplements and other therapies to treat these diseases.

This study involves research into the usefulness and safety of two probiotic products in maintaining remission in Crohn's disease and ulcerative colitis. Approximately 360 patients with Crohn's disease and ulcerative colitis from Ireland, Finland and Spain will be involved in the study. The yoghurts used in this study contain either Lactobacillus salivarius subsp. salivarius or Bifidobacterium infantis.

DETAILED DESCRIPTION:
There is a growing body of evidence that the enteric bacterial flora contribute to the pathogenesis of inflammatory bowel disease (IBD; Crohn's disease and Ulcerative Colitis) (Targan S and Shanahan F Inflammatory Bowel Disease: From Bench to Bedside, Williams and Wilkins 1994).

It has recently been found that patients suffering active Crohn's disease have significantly less recoverable bifidobacteria in their faeces compared to healthy individuals. This reduction in bifidobacteria numbers was observed to be directly correlated with decreased levels of B-D-galactosidase production and activity (Favier C et al. Dig Dis Sci 1997;42:817-822). B-D-galactosidase is an enzyme produced by bifidobacteria. These results support suggestions proposed in other studies (Bartram HP et al. Am J Clin Nutr 1994;59:428-432) that strains of bifidobacteria may play important roles in maintaining a balanced healthy intestinal microflora.

In Crohn's disease, there is extensive clinical evidence indicating the importance of the continuity of the faecal stream in disease recurrence.

Ingestion of bifidobacteria can improve gastrointestinal transit. In elderly individuals, mild constipation can be at least partially corrected through the consumption of milk fermented by bifidobacteria (Seki M et al. Nutr Food 1978;4:379-387). In addition, colonic transit times of women were significantly accelerated in the sigmoid colon following consumption of a milk fermented by bifidobacteria sp. and yoghurt cultures (Grimaud JC et al. Gastroenterol Clin Biol 1993;17:A127), but not by traditional yoghurt cultures alone (Grimaud JC et al. Les bact_ries lactiques, 1994;406).

Several genetically engineered 'knock out' and transgenic animal models of IBD have been reported in which the role of the enteric flora has been directly demonstrated by comparing animals raised in germ free versus conventional facilities. For example, the gastrointestinal Crohn's-like inflammation that occurs in interleukin-10 (IL-10) deficient mice is attenuated when the animals are kept in a germ free environment and becomes more pronounced and widespread when they are switched to conventional facilities. (Kuhn R et al. Cell 1993;75:263-274).

The mucosal inflammation in IL-10 deficient mice has been reported to be reduced by feeding the animals a preparation of lactobacilli (Madsen K et al Gastroenterology 1997;112:A1030), a result subsequently confirmed by a UCC-based research group who also reported that consumption of Lactobacillus salivarius UCC118 reduced cancer incidence (O'Mahony et al.2001).

Studies completed in rats have demonstrated that ingestion of bifidobacteria can suppress aberrant crypt foci (early preneoplastic lesions) formation in the colon (Kulkarni N and Reddy B. Proc Soc Experim Biol Med 1994;207:278-283) in addition to significant decreases in colon tumor incidence and in the numbers of tumors present (Singh J et al. Carcinogenesis 1997;18:833-841).

Background and Preliminary data:

Several probiotic strains of lactic acid bacteria and Bifidobacterium probiotic strains have been developed in UCC.

Lactobacillus salivarius UCC118 was chosen for its probiotic potential based on in vitro activity against several pathogens and several other properties including acid/bile tolerance. In addition, a preliminary trial, approved by the UCC Ethics Committee has already been conducted in 80 human volunteers and has shown that either milk or yoghurt may be used as a vehicle for delivery of Lactobacillus salivarius UCC118 to the gastrointestinal tract with equal efficacy in altering gut flora and apparent colonisation. An abstract, based on this study has been submitted to the American Gastroenterological Association and a full manuscript has been submitted for publication.

Furthermore, administration of Lactobacillus UCC118 to 20 patients with relapsed Crohn's disease over a six week period resulted in reports that consumption of the probiotic improved patient quality of life and, in fact, in most cases patients avoided the requirement for steroid use (McCarthy et al., Submitted).

Bifidobacterium infantis 35624 was chosen for its probiotic potential based on several physiological properties including acid/bile tolerance. In addition, preliminary trials completed by the UCC probiotic research group, in collaboration with UCLA School of Medicine (Division of Digestive Diseases), have shown that Bifidobacterium infantis 35624 or a combination of Lactobacillus salivarius UCC118 and Bifidobacterium infantis 35624 may prove more effective in beneficially altering gut flora in an inflammatory disease mouse model and of alleviating the symptoms of IBD in colonised mice. An abstract, based on this study has been submitted to the American Gastroenterological Association and a full manuscript is in preparation.

The primary aim of the study is to determine whether ingestion of probiotic preparations (containing Lactobacillus salivarius subsp. salivarius UCC118 or Bifidobacterium infantis 35624) can help in the maintenance of remission of patients with Crohn's disease and ulcerative colitis over a period of one year (i.e., delay the onset of relapse).

Secondary aims include an evaluation of the immunological and biochemical parameters of the immuno-inflammatory response and an assessment of the faecal flora in patients consuming the probiotic and control products.

ELIGIBILITY:
Inclusion Criteria for Crohn's Disease:

* Patients must be in clinical relapse with a CDAI score >150.
* Probiotic consumption must start within 2 weeks of commencing steroid use.
* To achieve remission, administration of steroids to the patients must follow the guidelines: Start dose of 40 mg per day, Taper daily dose by 5 mg per week every 1-2 weeks from 40 mg to 20 mg. Reduce thereafter from 20 mg - 0 mg ensuring the dosage is reduced to 0 mg by end of week 12.
* Patients must be taking 5-ASA.

Inclusion Criteria for Ulcerative Colitis:

* Patients must be within one month of entering remission following a documented episode of relapse (despite the use of 5-ASA).
* Remission is defined as patients who experience <3 bowel movements (without frank/gross blood) per day on >3 days out of 7 and are off all steroids including topical steroids.
* Patients may be receiving treatment involving 5-ASA or 5-ASP. However, this dose may not vary during the study.

Exclusion Criteria:

* Age - patients over 75 years will be excluded.
* Be pregnant, or have the desire to become pregnant during the study period.
* Patients with clinically significant immunodeficiency (quantitative immunoglobulin levels will be performed before entry to trial).
* Patients who are considered to be poor clinical attendees or be unlikely for any reason to be able to comply with the trial.
* Concomitant Drug usage - Patients may not be receiving any treatment with 6-Mercaptopurine, Azothioprine or cyclosporin.
* Patients may not be receiving treatment involving experimental drugs.
* Patients who have been on antibiotics within the previous month or who are likely to require antibiotics during the trial period will be excluded.
* Previous surgery - patients will be excluded if the have undergone resection of more than one (1) metre of bowel in the past. Patients who have undergone less extensive surgical resection of bowel will be eligible provided there is objective (endoscopic or radiological) evidence of recurrence.
* Malignancy or any concomitant end-stage organ disease.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2002-01; Study Completion 2007-11

PRIMARY OUTCOMES:
To determine whether ingestion of probiotic preparations (containing Lactobacillus salivarius subsp. salivarius UCC118 or Bifidobacterium infantis 35624) can help in the maintenance of remission of patients with Crohn's disease and ulcerative colitis | One year

SECONDARY OUTCOMES:
Evaluation of the immunological and biochemical parameters of the immuno-inflammatory response and an assessment of the faecal flora in patients consuming the probiotic and control products | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Fergus Shanahan, Prof, Principal Investigator — Cork University Hospital & University College Cork
Locations (1):
- Cork University Hospital, Cork, Co Cork, Ireland

REFERENCES:
- See also: Related Info — http://apc.ucc.ie